CLINICAL TRIAL: NCT00162279
Title: A Multi-Center, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety and Clinical Efficacy of Intravenous Infusions of BMS-188667 (10 mg/kg) Given Monthly in Combination With Subcutaneous Injections of Etanercept (25mg)Given Twice Weekly to Subjects With Active Rheumatoid Arthritis
Brief Title: The Study of Abatacept in Combination With Etanercept
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-101
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

INTERVENTIONS:
Drug: Abatacept

SUMMARY:
The Study was designed to look at the safety and efficacy of abatacept in combination with etanercept.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who had completed the short term portion of IM101-101.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141
Dates: Start 2000-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Abatacept combined with etanercept will have greater clinical efficacy compared to subjects receiving etanercept alone | at 6 months

SECONDARY OUTCOMES:
ACR 50 and 70 will be evaluated | at 6 months

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Local Institution, Huntsville, Alabama
  - Local Institution, La Jolla, California
  - Local Institution, Long Beach, California
  - Local Institution, Los Angeles, California
  - Local Institution, Palo Alto, California
  - Local Institution, San Francisco, California
  - Local Institution, Denver, Colorado
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Titusville, Florida
  - Local Institution, Rome, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Hagerstown, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Duluth, Minnesota
  - Local Institution, Lincoln, Nebraska
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, Los Alamos, New Mexico
  - Local Institution, Albany, New York
  - Local Institution, Mineola, New York
  - Local Institution, New York, New York
  - Local Institution, Bismarck, North Dakota
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Duncansville, Pennsylvania
  - Local Institution, Norristown, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Knoxville, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Temple, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Edmonds, Washington
  - Local Institution, Tacoma, Washington
  - Local Institution, Glendale, Wisconsin